CLINICAL TRIAL: NCT01843894
Title: A Phase 1/2, First-in-Human, Double-Masked, Placebo-Controlled, Dose-Escalation Study Evaluating the Safety, Tolerability, and Efficacy of RU-101 Ophthalmic Solution in Patients With Severe Dry Eye
Brief Title: A Phase 1/2, RU-101 Ophthalmic Solution in Patients With Severe Dry Eye
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: R-Tech Ueno, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: RU-101-C001
Record Dates: First submitted 2013-04-12; First posted 2013-05-01 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Dry Eye
Keywords: sever dry eye,keratoconjunctivitis sicca
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Ruthenium-101

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): In Stage I, each patient will instill 1 drop of placebo into each eye, 6 times a day with at least 2 hours between each dose, for 28 days (4 weeks; a total of 168 doses to each eye). In Stage II, each patient will instill 1 drop into each eye, 6 times a day with at least 2 hours between each dose, for 84 days (12 weeks; a total of 504 doses to each eye).
  Interventions: Biological: RU-101
- RU-101 (Experimental): In Stage I, each patient will instill 1 drop of RU-101 ophthalmic solution (5%, 10%, or 15%) into each eye, 6 times a day with at least 2 hours between each dose, for 28 days (4 weeks; a total of 168 doses to each eye). In Stage II, each patient will instill 1 drop of RU-101 ophthalmic solution (selected dose from Stage I) into each eye, 6 times a day with at least 2 hours between each dose, for 84 days (12 weeks; a total of 504 doses to each eye).
  Interventions: Biological: RU-101

INTERVENTIONS:
Biological: RU-101 — Recombinant human serum albumin

SUMMARY:
Objectives:

Primary

* To determine the safety and tolerability of escalating doses of RU-101 for 4 weeks in patients with severe dry eye

Secondary

* To explore the efficacy of RU-101
* To explore optimal endpoints for future studies

DETAILED DESCRIPTION:
This is a Phase 1/2, first-in-human, multicenter, dose escalation, double-masked, placebo controlled study consisting of two stages. In Stage I, 3 cohorts are planned to evaluate escalating doses of RU 101 ophthalmic solution, instilled 6 times daily into each eye for 4 weeks (28 days). Each cohort will comprise 4 patients randomized 3:1 to RU-101 or placebo. A masked safety data review will be performed prior to each dose escalation to determine if any dose limiting toxicities (DLTs) occurred and to define the MTD or highest dose to be used in Stage II. In Stage II, an expanded cohort will receive the dose defined in Stage I (MTD or highest dose if MTD is not reached), instilled 6 times daily into each eye for 12 weeks (84 days). The expanded cohort will comprise approximately 96 patients randomized 1:1 to RU-101 or placebo, provided in a double-masked manner.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 to 80 years.
2. Patients have had dry eye symptoms at least 4 months.
3. Patients have the following signs in the worst eye:

   1. Corneal staining score with fluorescein staining ≥ 6/15 with at least one in the central
   2. Conjunctival staining score with Lissamine Green ≥ 2/18
4. Patients who had been receiving treatment with eye drops of artificial tears, Restasis, or topical steroids but have had insufficient efficacy or have found these products to be intolerable. If using Restasis or topical steroids, patients must agree to a 30-day washout period prior to the first IP dose (Day 0).
5. Female patients of child bearing potential must agree to have a urine pregnancy test performed at Screening (must be negative) and agree to use a medically acceptable form of birth control (e.g., intrauterine device, birth control pill, patch or subcutaneous implant, condoms, diaphragm, or abstinence) throughout the duration of IP instillation. Women considered capable of becoming pregnant include all females who have experienced menarche and who have not experienced menopause (as defined by amenorrhea for > 12 consecutive months) or have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy).

Exclusion Criteria:

1. Presence of anterior eye diseases except dry eye.
2. Intraocular pressure ≥ 22 mmHg at Screening.
3. Use of any ophthalmic solutions (including over-the-counter [OTC] solutions), serum eye drops, or contact lenses during the Treatment Phase. Artificial tears are allowed during the Screening Phase but must not be used from the first dose (Day 0) through the Treatment Phase.
4. Use of eye drops of Restasis or topical steroids within 30 days of the first dose (Day 0).
5. Use of antihistamines, beta blockers, tricyclic antidepressants, or antidepressants with anticholinergic side effects during the Treatment Phase.
6. Patients with previous corneal transplantation or laser-assisted in situ keratomileusis (LASIK).
7. Presence of graft-versus-host disease (GVHD).
8. Patients who have had other ocular surgery within 3 months prior to the first dose.
9. Patients with punctal plugs or punctal cautery < 3 months prior to the first dose.
10. Patients with severe dry eye due to Stevens-Johnson disease or ocular cicatricial pemphigoid.
11. History of allergy to human serum protein products and/or any history of allergy to yeast.
12. History of allergies to recombinant products, ophthalmic solutions, any constituents of RU 101, or any solutions planned for use in this study.
13. Any significant chronic illness that, in the opinion of the Principal Investigator (PI), could interfere with the study parameters.
14. Use of any investigational product or device within 30 days prior to the Screening Visit or during the study.
15. Known history of alcohol and/or drug abuse within the past 12 months, which in the opinion of the PI could interfere with study compliance, outcome measures including safety parameters, and/or the general medical condition of the patient.
16. Those unable in the opinion of the PI to comply fully with the study requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Occular Adverse Events | 56 dyas (stage1) 112 days (stage 2)
  The number of participants with a change from baseline in the following symptoms:
  * intraocular pressure (IOP)-The IOP assessment will be done using either a Goldmann applanation tonometer or digital tonometer.
  * slit lamp biomicroscopy
  * fundoscopy-A dilated fundoscopic examination including evaluation of the vitreous, optic nerve, macula and retina will be performed and any abnormalities will be evaluated on a 4-point scale (1-4; slight, moderate, severe, or very severe

SECONDARY OUTCOMES:
Symptoms | 28days (stage 1) 3 months (stage2)
  The number of participants with a change from baseline in the following symptoms:
  * Symptom Assessment in Dry Eye (SANDE)
  * Ocular Surface Disease Index (OSDI)
  * Visual acuity (Early Treatment Diabetic Retinopathy Study [ETDRS] chart, high and 10% low contrast)
Signs | 28days (stage 1) 3 months (stage2)
  The number of participants with a change from baseline in the following signs:
  * Tear break-up time (TBUT)
  * Corneal staining with fluorescein
  * Conjunctival staining with Lissamine Green
  * Corneal sensitivity
  * Schirmer test
Non-Occular Adverse Events | 56 dyas (stage1) 112 days (stage 2)
  Number of AEs will be measured (vital signs, physical examination results, safety laboratory results, 12-lead electrocardiogram (ECG), and IP comfort assessment.

CONTACTS AND LOCATIONS:
Overall Officials: John Sheppard, MD, Principal Investigator — Virginia Ehe Consultants
Locations (1):
- Virginia Eye Consultants, Norfolk, Virginia, United States